CLINICAL TRIAL: NCT01239563
Title: THYMOGLOBULIN INDUCTION AND STEROID-FREE IMMUNOSUPPRESSION IN KIDNEY TRANSPLANTATION FROM DECEASED DONORS AFTER CARDIAC DEATH-AN OPEN LABEL RANDOMISED CONTROLLED TRIAL TO EVALUATE THE ROLE OF THYMOGLOBULIN AS INDUCTION IMMUNOSUPPRESSION IN KIDNEY TRANSPLANTS FROM DECEASED DONORS AFTER CARDIAC DEATH
Brief Title: Thymoglobulin Induction in Kidney Transplant Recipients
Acronym: TIKT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Peter Friend / Professor of Transplantation, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oxford/OTC/TIKT; 2009-016676-73 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Kidney Transplantation; Ischemia-Reperfusion Injury
Keywords: kidney transplantation; donation after cardiac death; ischemia-reperfusion injury; thymoglobulin; steroid avoidance; lymphocyte
MeSH Terms: conditions — Reperfusion Injury | interventions — Antilymphocyte Serum; thymoglobulin; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymoglobulin (Experimental): Thymoglobulin induction group
  Interventions: Drug: antithymocyte globulin
- Basiliximab (Active Comparator): Basiliximab induction - 20 mg, day 0 and day 4
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: antithymocyte globulin — Thymoglobulin 1.5mg/kg, 4 doses Thymoglobulin 6mg/kg, single dose
  Other Names: Thymoglobulin, L04AA04
  Arms: Thymoglobulin
Drug: Basiliximab — Intravenous 20mg, day 0&4
  Other Names: Simulect
  Arms: Basiliximab

SUMMARY:
The purpose of this study is to determine if anti-thymocyte globulin (Thymoglobuline) administration in the kidney transplant recipient is able to reduce the amount of damage that kidneys transplanted from deceased donors sustains on reperfusion.

DETAILED DESCRIPTION:
The increasing disparity between organ availability and the number of patients on waiting list for a transplant has led to different strategies to improve half life of all transplants. One such method is to reduce the amount of damage the organ sustains during the period of preservation and reperfusion in the recipient. Thymoglobulin, an anti-lymphocyte antibody has been shown to have the ability to reduce this damage in experimental studies. This study aims to ascertain the role of Thymoglobulin in kidney transplants from donors after cardiac death, the type of kidney transplants at highest risk of sustaining injury during preservation. The study will involve comparison with conventional immunosuppressant therapy, comparison between Thymoglobulin administered in different doses, and observation of the patterns of blood cell repopulation (lymphocytes mainly) in the first year following kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* Recipient of DCD kidney transplant
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the first 12 months of the study
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:
* Failure of either recipient of a pair of kidneys to give consent
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* History of specific viral infection that would contraindicate depleting antibody therapy e.g. hepatitis B&C, HIV
* Significant hepatic impairment-.i.e. Values 3 times upper limit of normal (unless this is usual for the subject)
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Participants who have participated in another research study involving an investigational product in the previous 12 weeks
* Previous administration of Thymoglobuline
* Patients with functioning non-renal transplants and on immunosuppression
* The patient is not suitable, in the opinion of the Investigator, to take part in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
delayed graft function | 7 days

SECONDARY OUTCOMES:
steroid avoidance | 1 year
lymphocyte repopulation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Friend, MD FRCS, Principal Investigator — University of Oxford; Susan V Fuggle, DPhil MRCPath, Study Director — Oxford Radclifffe Hospitals NHS Trust; Kathryn Wood, DPhil BSc, Study Director — University of Oxford
Locations (2):
- United Kingdom (2):
  - Oxford Transplant Centre, Churchill Hospital, Oxford, Oxfordshire
  - University of Oxford, Oxford, Oxfordshire